CLINICAL TRIAL: NCT03607916
Title: Estimation of the Effective Dose (ED) 95 of Intrathecal Hyperbaric Prilocaine 2% for Scheduled Cesarean Delivery : a Dose-finding Study Based on the Continual Reassessment.
Brief Title: Estimation of the Effective Dose (ED) 95 of Intrathecal Hyperbaric Prilocaine 2% for Scheduled Cesarean Delivery.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B076201524085
Record Dates: First submitted 2018-07-24; First posted 2018-07-31 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Pregnant Women
Keywords: Scheduled cesarean delivery,spinal anesthesia,local anesthesia
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (10):
- Cohort 1 : HB Prilocaine 2%,(60mg) (Experimental): Dose-finding study with 4 subjects per dose and a maximum of 40 parturients.To identify the dose to give for reaching the ED95 (effective dose for 95% subjects), Hyperbaric prilocaine 2% will be administered at the dose initial of 60 mg in the cohort 1 (4 subjects), then the dose will be adjusted in the next cohorts using the Continual Reassessment Method (CRM). The dose range will be from 45 to 70mg.
  Interventions: Drug: Hyperbaric prilocaine 2%; Drug: Morphine
- Cohort 2 : HB Prilocaine 2%,(45-70mg) (Experimental): Dose-finding study with 4 subjects per dose and a maximum of 40 parturients.To identify the dose to give for reaching the ED95 (effective dose for 95% subjects), Hyperbaric prilocaine 2% will be administered at the dose initial of 60 mg in the cohort 1 (4 subjects), then the dose will be adjusted in the next cohorts using the Continual Reassessment Method (CRM). The dose range will be from 45 to 70mg.
  Interventions: Drug: Hyperbaric prilocaine 2%; Drug: Morphine
- Cohort 3 : HB Prilocaine 2%,(45-70mg) (Experimental): Dose-finding study with 4 subjects per dose and a maximum of 40 parturients.To identify the dose to give for reaching the ED95 (effective dose for 95% subjects), Hyperbaric prilocaine 2% will be administered at the dose initial of 60 mg in the cohort 1 (4 subjects), then the dose will be adjusted in the next cohorts using the Continual Reassessment Method (CRM). The dose range will be from 45 to 70mg.
  Interventions: Drug: Hyperbaric prilocaine 2%; Drug: Morphine
- Cohort 4 : HB Prilocaine 2%,(45-70mg) (Experimental): Dose-finding study with 4 subjects per dose and a maximum of 40 parturients.To identify the dose to give for reaching the ED95 (effective dose for 95% subjects), Hyperbaric prilocaine 2% will be administered at the dose initial of 60 mg in the cohort 1 (4 subjects), then the dose will be adjusted in the next cohorts using the Continual Reassessment Method (CRM). The dose range will be from 45 to 70mg.
  Interventions: Drug: Hyperbaric prilocaine 2%; Drug: Morphine
- Cohort 5 : HB Prilocaine 2%,(45-70mg) (Experimental): Dose-finding study with 4 subjects per dose and a maximum of 40 parturients.To identify the dose to give for reaching the ED95 (effective dose for 95% subjects), Hyperbaric prilocaine 2% will be administered at the dose initial of 60 mg in the cohort 1 (4 subjects), then the dose will be adjusted in the next cohorts using the Continual Reassessment Method (CRM). The dose range will be from 45 to 70mg.
  Interventions: Drug: Hyperbaric prilocaine 2%; Drug: Morphine
- Cohort 6 : HB Prilocaine 2%,(45-70mg) (Experimental): Dose-finding study with 4 subjects per dose and a maximum of 40 parturients.To identify the dose to give for reaching the ED95 (effective dose for 95% subjects), Hyperbaric prilocaine 2% will be administered at the dose initial of 60 mg in the cohort 1 (4 subjects), then the dose will be adjusted in the next cohorts using the Continual Reassessment Method (CRM). The dose range will be from 45 to 70mg.
  Interventions: Drug: Hyperbaric prilocaine 2%; Drug: Morphine
- Cohort 7 : HB Prilocaine 2%,(45-70mg) (Experimental): Dose-finding study with 4 subjects per dose and a maximum of 40 paturients.To identify the dose to give for reaching the ED95 (effective dose for 95% subjects), Hyperbaric prilocaine 2% will be adminitrated at the dose initial of 60 mg in the cohort 1 (4 subjects), then the dose will be adjusted in the next cohorts using the Continual Reassessment Method (CRM). The dose range will be from 45 to 70mg.
  Interventions: Drug: Hyperbaric prilocaine 2%; Drug: Morphine
- Cohort 8 : HB Prilocaïne 2%,(45-70mg) (Experimental): Dose-finding study with 4 subjects per dose and a maximum of 40 parturients.To identify the dose to give for reaching the ED95 (effective dose for 95% subjects), Hyperbaric prilocaine 2% will be administered at the dose initial of 60 mg in the cohort 1 (4 subjects), then the dose will be adjusted in the next cohorts using the Continual Reassessment Method (CRM). The dose range will be from 45 to 70mg.
  Interventions: Drug: Hyperbaric prilocaine 2%; Drug: Morphine
- Cohort 9 : HB Prilocaine 2%,(45-70mg) (Experimental): Dose-finding study with 4 subjects per dose and a maximum of 40 parturients.To identify the dose to give for reaching the ED95 (effective dose for 95% subjects), Hyperbaric prilocaine 2% will be administered at the dose initial of 60 mg in the cohort 1 (4 subjects), then the dose will be adjusted in the next cohorts using the Continual Reassessment Method (CRM). The dose range will be from 45 to 70mg.
  Interventions: Drug: Hyperbaric prilocaine 2%; Drug: Morphine
- Cohort 10 : HB Prilocaine 2%,(45-70mg) (Experimental): Dose-finding study with 4 subjects per dose and a maximum of 40 parturients.To identify the dose to give for reaching the ED95 (effective dose for 95% subjects), Hyperbaric prilocaine 2% will be administered at the dose initial of 60 mg in the cohort 1 (4 subjects), then the dose will be adjusted in the next cohorts using the Continual Reassessment Method (CRM). The dose range will be from 45 to 70mg.
  Interventions: Drug: Hyperbaric prilocaine 2%; Drug: Morphine

INTERVENTIONS:
Drug: Hyperbaric prilocaine 2% — Varying dose according to sensitive response of previous subjects. All study doses of hyperbaric prilocaine 2% will be administrated intrathecally with 100µg of morphine
  Other Names: Tachipri
  Arms: Cohort 10 : HB Prilocaine 2%,(45-70mg); Cohort 2 : HB Prilocaine 2%,(45-70mg); Cohort 3 : HB Prilocaine 2%,(45-70mg); Cohort 4 : HB Prilocaine 2%,(45-70mg); Cohort 5 : HB Prilocaine 2%,(45-70mg); Cohort 6 : HB Prilocaine 2%,(45-70mg); Cohort 7 : HB Prilocaine 2%,(45-70mg); Cohort 8 : HB Prilocaïne 2%,(45-70mg); Cohort 9 : HB Prilocaine 2%,(45-70mg)
Drug: Hyperbaric prilocaine 2% — The dose of 60 mg of Hyperbaric prilocaine 2% will be administrated intrathecally with 100µg of morphine
  Other Names: Tachipri
  Arms: Cohort 1 : HB Prilocaine 2%,(60mg)
Drug: Morphine — 100µg morphine

SUMMARY:
Prilocaine is a local anesthetic drug which as an intermediate duration of action shorter than bupivacaine 0,5% that is usually used for spinal anesthesia in scheduled cesarean section. No study has yet investigated the use of hyperbaric (HB) prilocaine 2% for intrathecal anesthesia in cesarean section. The aim of this study is to determine the Effective Dose (ED) 95 of hyperbaric (HB) prilocaine 2% by using the Continual Reassessment Method (CRM)

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status (ASA) < III
* Age 18-40 year
* Body Weight <100 kg
* Height between 160 and 175 cm
* Gestational age>37 SA
* Elective cesarean delivery
* Singleton pregnancy
* Non complicated pregnancy
* Signed informed consent obtained prior to any study specific assessments and procedures

Exclusion Criteria:

* Twin pregnancy
* History of 2 cesarean section or more
* Diabetes and gestational diabetes
* Placenta praevia
* Congenital foetal abnormality
* Patient in labour
* Membrane rupture
* Known allergy to local anaesthetics
* Disagreement of the patient
* Pregnancy-induced hypertension
* Pre eclampsia and eclampsia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Success of anesthesia | during surgery (average 1 hour)
  The nerve blockade will be considered as success when a bilateral T4 level will reach in 15 minutes after intrathecal injection without additional epidural injection needed within 45 minutes peri-operative ; no pain at the skin incision, no pain during 45 minutes after the skin incision

SECONDARY OUTCOMES:
Level of Sensory block assessed as loss of sensation to pinprick, cold and pressure | Until complete release of sensory block (T12-S1) (average 4 hours)
  Every 2 minutes after spinal anesthesia during 15 minutes, then every 5 minutes until the end of surgery, thereafter, once every hour until total regression of sensory block (T12-S1).
Side-effects (nausea, vomiting,pruritus) | up to 24 hours after surgery
  from 15 minutes after spinal anesthesia and every 4 hours for 24 hours (score 0=no symptoms; 1=symptoms with no treatment necessary; 2=symptoms present and treated)
Transient neurologic symptoms (TNS) | up to 5 Days
  TNS are defined as pain and/or dysesthesia occured after complete release of sensory block at the gluteal level, at the tights and at the legs. At Day 0, Day 1, day 3 and Day 5
Pain as assessed by Visual Analogue Scale (VAS) | during surgery (average 1 hour)
  Pain levels will be determined every 5 minutes during surgery. The Visual Analogue score (scale : 0 = no pain; 10= worst pain imaginable)
Number of participants with low blood pressure | during surgery (average 1 hour)
  Arterial blood pressure will be measured at every 2.5 minute during the first 15 minutes, then at every 5 minutes until the end of surgery. A blood pressure lower is define as a blood pressure lower than 20% or more than the basal blood pressure (Systolic blood pressure before spinal anesthesia)
Methemoglobinemia | at delivery (average 1 hour)
  Methemoglobin level measured in umbilical cord blood of new born at the delivery

CONTACTS AND LOCATIONS:
Overall Officials: Panayota KAPESSIDOU, MD, PhD, Study Director — University Hospital Saint-Pierre (CHU Saint-Pierre), Université Libre de Bruxelles (ULB); Philippe Goffard, MD, Principal Investigator — University Hospital Saint-Pierre (CHU Saint-Pierre), Université Libre de Bruxelles (ULB)
Locations (1):
- University Hospital Saint-Pierre, Université Libre de Bruxelles, Brussels Capital Region, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Camponovo C, Fanelli A, Ghisi D, Cristina D, Fanelli G. A prospective, double-blinded, randomized, clinical trial comparing the efficacy of 40 mg and 60 mg hyperbaric 2% prilocaine versus 60 mg plain 2% prilocaine for intrathecal anesthesia in ambulatory surgery. Anesth Analg. 2010 Aug;111(2):568-72. doi: 10.1213/ANE.0b013e3181e30bb8. Epub 2010 Jun 7. PMID 20529983
- [Background] Gupta PK, Chevret S, Zohar S, Hopkins PM. What is the ED95 of prilocaine for femoral nerve block using ultrasound? Br J Anaesth. 2013 May;110(5):831-6. doi: 10.1093/bja/aes503. Epub 2013 Feb 7. PMID 23393153